CLINICAL TRIAL: NCT01480856
Title: Evaluation of the Efficacy of Cobedding in Daily Weight Gain of Neonate Twins
Brief Title: Cobedding in Daily Weight Gain of Neonate Twins
Acronym: Cobedding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08/2-H
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Preterm Newborn Twins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cobedding (Active Comparator): Newborn twins are settled in a single bed : this is cobedding
  Interventions: Procedure: Cobedding
- Single -bedding (Placebo Comparator): Newborn twins are settled in two beds : this is single-bedding
  Interventions: Procedure: Single-bedding

INTERVENTIONS:
Procedure: Cobedding — Newborn twins are settled in a singe bed: this is cobedding
  Arms: Cobedding
Procedure: Single-bedding — Newborn twins are settled in two single beds : this is single-bedding
  Arms: Single -bedding

SUMMARY:
Cobedding consists of associating twins in a common cocoon in order to maintain links developed in utero and reduce the stress of premature birth. The aim of this randomized, controlled prospective study is to compare efficacy (in term of newborn daily weight gain) and safety of cobedding versus single-bedding of preterm twins.

DETAILED DESCRIPTION:
Randomization will occur during the first 96 hours after birth.Twins randomized in the cobedding arm will be kept in the same cocoon until maximum 37 amenorrhea weeks. Each day, parameters (weight gain, …) will be registered.At two years old, neuromotor development of twins will be estimated by Brunet-Lezine test.

ELIGIBILITY:
Inclusion Criteria:

* At time of inclusion, twins must have been separated since less than 96h following birth.
* twins born between 30 to 34 weeks of gestation
* no severe congenital pathology
* hospitalized at the intensive neonates care unit
* Parents having given their non-opposition to this study within the 96 hours following twins birth -Time length of cobedding estimated by the investigator to be of three weeks -

Exclusion Criteria:

Inclusion criteria not fulfilled

* safety reasons
* prolonged lack of comfort clinically harmful for the newborn as per investigator conclusion.

Max Age: 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2012-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Daily weight gain of cobedded preterm twins versus that of single-bedded preterm twins | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  The main objective of this study is to compare daily weight gain of cobedded preterm twins versus that of single-bedded preterm twins

SECONDARY OUTCOMES:
cardiorespiratory stability | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  cardiorespiratory stability
Thermoregulation | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  Thermoregulation
parents well-being estimated through questionnaires | 5 weeks
  parents well-being estimated through questionnaires
newborns comfort | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  newborns comfort
stop date of parenteral nutrition | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  stop date of parenteral nutrition
date of removal of central catheter | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  date of removal of central catheter
date of removal of nasogastric catheter | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  date of removal of nasogastric catheter
stop date of oxygenotherapy | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  stop date of oxygenotherapy
neuromotor development estimated by "Brunet Lezine" test at 2 years old | 2 years
  neuromotor development estimated by "Brunet Lezine" test at 2 years old
Hospitalization time length | patients will be followed for the duration of hospital stay in special bed (cobedding or single bed) , an expected average of 5 weeks
  Hospitalization time length

CONTACTS AND LOCATIONS:
Locations (1):
- Universitary Hospital Center, Nantes, Loire atlantique, France